CLINICAL TRIAL: NCT04859335
Title: Prospective Study : Long-term Evolution of Balance and Vestibular Function in Patients Treated With Gammaknife Radiosurgery for Vestibular Schwannoma EQUI-GAMMA
Brief Title: Evolution of Balance and Vestibular Function in Patients Treated With Gammaknife Radiosurgery for Vestibular Schwannoma
Acronym: EQUI-GAMMA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: RC31/21/0034
Record Dates: First submitted 2021-04-16; First posted 2021-04-26 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-08

CONDITIONS: Vestibular Schwannoma
Keywords: Vestibular Schwannoma; Gammaknife radiosurgery; Dizziness; Balance
MeSH Terms: conditions — Neuroma, Acoustic; Dizziness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Schwannomas patients needing gammaknife radiosurgery (Other): Patients will undergo balance and hearing questionnaires before and after gammaknife radiosurgery.
  This is a before/after analysis needing only one arm: the "before" data will serve as control to the "after" data
  Interventions: Radiation: gammaknife radiosurgery

INTERVENTIONS:
Radiation: gammaknife radiosurgery — Patients will undergo questionnaires before the gammaknife radiosurgery, then one year and three years after the intervention.

SUMMARY:
Vestibular schwannomas are benign lesions of the ponto-cerebellar angle that are potentially dangerous because of their growth in a cramped space and the compressive phenomena they can cause. Stereotactic Gammaknife radiosurgery is a treatment option that can be offered for evolutive schwannomas smaller than 2.5-3 cm in size. It allows tumor stabilisation in 85% of cases with less than 1% facial nerve damage risk.

There are controversial results regarding hearing preservation : percentages vary between 25 and 80% in the literature, depending on the criteria used and the post-treatment delay.

Few studies have investigated changes in vestibular function and the impact on balance of radiosurgery, and their results are variable.

These controversial results lead us to comprehensively assess the vestibular function and balance of these patients using a balance-specific quality of life questionnaire, in addition to objective overall vestibular assessments of vestibular function.

DETAILED DESCRIPTION:
Vestibular schwannomas are benign lesions of the ponto-cerebellar angle that are potentially dangerous because of their growth in a cramped space and the compressive phenomena they can cause. Stereotactic Gammaknife radiosurgery is a treatment option that can be offered for evolutive schwannomas smaller than 2.5-3 cm in size. It allows tumor stabilisation in 85% of cases with less than 1% facial nerve damage risk.

There are controversial results regarding hearing preservation : percentages vary between 25 and 80% in the literature, depending on the criteria used and the post-treatment delay.

Few studies have investigated changes in vestibular function and the impact on balance of radiosurgery.Their results are heterogeneous, on one hand, indicating little worsening of symptoms, or even improvement in some studies. On the other hand, a 2017 study reported symptomatic worsening of caloric response deficits in 17.6% of cases. Vestibular function at high frequencies or for otolithic organs (utricle and saccule) has hardly ever been explored.

The largest cohort, reported in "gammaknife radiosurgery for vestibular schwannomas a quality of life evaluation" concerns 353 patients and shows that the overall quality of life of the patients treated is on average comparable to that of the general population but that the vertigo is more frequent in this population, with a more marked impact on the overall quality of life.

These controversial results lead us to comprehensively assess the vestibular function and balance of these patients using a balance-specific quality of life questionnaire, in addition to objective overall vestibular assessments of vestibular function.

Thus, the present study aims to assess the quality of balance of patients treated with Gammaknife radiosurgery for vestibular schwannoma at 1 year and 3 years after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Vestibular schwannoma's Patients for whom an indication of gammaknife radiosurgery was determined in a dedicated multidisciplinary consultation meeting, having not received previous treatment for this schwannoma.
* Patient affiliated to Social Security
* No opposition to participation

Exclusion Criteria:

* History of prior treatment for the presented vestibular schwannoma (surgery, fractional radiotherapy)
* History of otological or otoneurological pathology associated with schwannoma
* Patient with type 2 neurofibromatosis
* Patient under legal protection
* Pregnant or breastfeeding women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-05-21 (Actual); Primary Completion 2028-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
quality of the perceived balance, assessed by the French version of the Dizziness Handicap Inventory (DHI) | before gamma knife radiosurgery (Baseline)
  Questionnaire including 25 items with a "yes/no/maybe" answer possibility
quality of the perceived balance, assessed by the French version of the Dizziness Handicap Inventory (DHI) | One year after gamma knife radiosurgery
  Questionnaire including 25 items with a "yes/no/maybe" answer possibility
quality of the perceived balance, assessed by the French version of the Dizziness Handicap Inventory (DHI) | Three years after gamma knife radiosurgery
  Questionnaire including 25 items with a "yes/no/maybe" answer possibility

SECONDARY OUTCOMES:
Evolution of hearing | before gamma knife radiosurgery (Baseline)
  Evaluate the evolution of hearing using data obtained during tonal audiometry (frequency by frequency between 250 Hz and 8 kHz, average hearing loss calculated on the frequencies 0.5, 1, 2, and 4 kHz)
Evolution of hearing | One year after gamma knife radiosurgery
  Evaluate the evolution of hearing using data obtained during tonal audiometry (frequency by frequency between 250 Hz and 8 kHz, average hearing loss calculated on the frequencies 0.5, 1, 2, and 4 kHz)
Evolution of hearing | Three years after gamma knife radiosurgery
  Evaluate the evolution of hearing using data obtained during tonal audiometry (frequency by frequency between 250 Hz and 8 kHz, average hearing loss calculated on the frequencies 0.5, 1, 2, and 4 kHz)

CONTACTS AND LOCATIONS:
Overall Officials: Mathieu MARX, MD PhD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- CHU Toulouse, Toulouse, France